CLINICAL TRIAL: NCT01903811
Title: A Phase II Randomized Study Comparing Two Doses of Carfilzomib (NSC-756640) With Dexamethasone for Multiple Myeloma Patients With Relapsed or Refractory Disease
Brief Title: S1304, Carfilzomib and Dexamethasone for Treating Patients With Relapsed or Refractory Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: S1304; NCI-2013-00796 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PS1304_A07PAMDREVW01; SWOG-S1304; S1304 (Other: SWOG); S1304 (Other: CTEP); U10CA180888 (NIH); U10CA032102 (NIH)
Record Dates: First submitted 2013-07-16; First posted 2013-07-19 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
Keywords: carfilzomib; relapsed; refractory; multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (dexamethasone, low-dose carfilzomib) (Experimental): Patients receive dexamethasone IV and low-dose carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16. (Note that course 1 is given at a reduced dose.) Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients with progression cross-over to Arm II.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis
- Arm II (dexamethasone, high-dose carfilzomib) (Experimental): Patients receive dexamethasone IV and high-dose carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16. (Note that course 1 is given at a reduced dose over 2-10 minutes.) Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: Dexamethasone — Given IV
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial compares how well two different doses of carfilzomib work when given with dexamethasone in treating patients with multiple myeloma that has come back after a period of improvement or has not responded to treatment. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving carfilzomib together with dexamethasone may kill more cancer cells. It is not yet known whether a higher or lower dose of carfilzomib works better when given with dexamethasone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate and compare progression free survival (PFS) of two different doses of carfilzomib with dexamethasone in multiple myeloma (MM) patients with relapsed and/or refractory disease.

SECONDARY OBJECTIVES:

I. To evaluate and compare response rates (RR) for each arm. II. To evaluate response rates (RR) for patients that relapse on low dose carfilzomib and subsequently cross-over to high dose carfilzomib.

III. To evaluate the safety of this combination for this patient population. IV. To evaluate overall survival (OS).

TERTIARY OBJECTIVES:

I. To explore the molecular variability in MM cells obtained from extramedullary bone marrow relapse sites.

II. To explore the role of positron emission tomography (PET) scanning in assessing disease burden and as a tool to assess treatment response.

III. To explore changes in left ventricular ejection fraction (LVEF) in patients with relapsed or refractory multiple myeloma treated with low dose carfilzomib or high dose carfilzomib plus dexamethasone.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive dexamethasone intravenously (IV) and low-dose carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16. Patients with progression cross-over to Arm II.

ARM II: Patients receive dexamethasone IV and high-dose carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16.

Note that for the first course of treatment on both arms carfilzomib is given at a reduced rate to assess toxicity.

In both arms, treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 3 years from initial registration.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION STEP 1: INITIAL RANDOMIZATION
* Patients must have a confirmed diagnosis of symptomatic multiple myeloma and must be currently relapsed or refractory; all tests for establishing disease status must be completed within 28 days prior to registration and documented on the Baseline Tumor Assessment Form for Multiple Myeloma
* Patients must have measurable disease within 28 days prior to registration
* Patients must have received at least one prior regimen of chemotherapy for symptomatic multiple myeloma; patients may not have more than six (6) previous regimens of therapy for the disease; prior chemotherapy must have been completed at least 21 days prior to registration; for study purposes, a regimen is defined as follows:

  * An anti-myeloma therapy used at the time of initial diagnosis or documented disease progression which is given with the intent to decrease disease burden
  * Any maintenance therapy used after an Induction should be considered part of that Induction regimen
  * Use of any agent or combination of agents more than once during the patient's disease history for separate documented disease progressions will be counted as separate regimens (e.g., if a patient receives lenalidomide/bortezomib at initial diagnosis and achieves response, but then progresses and receives lenalidomide/bortezomib after progression, these count as 2 separate regimens)
  * In cases of allogeneic or autologous stem cell transplant, the entire induction + stem cell mobilization + conditioning + planned maintenance should be considered one regimen
* Patients may not have received any prior carfilzomib treatment
* Patients must not be receiving any other concurrent therapy considered to be investigational; patients must not be planning to receive any radiotherapy (except localized radiation for palliative care); patients must not be planning to receive any concurrent chemotherapy, immunotherapy, radiotherapy or other treatment with curative intent
* Patients must have complete history and physical examination within 28 days prior to registration
* Patients must have baseline PET scan within 28 days prior to registration; note that images are submitted centrally for review
* Patients with non-secretory MM or known primary amyloidosis are not eligible
* Patients must have Zubrod performance status 0-2
* Patients must not have clinically significant illness including uncontrolled, active infection requiring intravenous antibiotics, New York Heart Association (NYHA) class III or class IV heart failure, unstable angina pectoris, myocardial infarction within the past 6 months, or >= grade 3 cardiac arrhythmias
* Patients must have undergone an electrocardiogram (EKG) within 28 days prior to registration
* Patients must have either echocardiogram (ECHO) with ejection fraction >= 45% within 28 days prior to registration
* Patients must not have > grade 2 neuropathy and/or POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum glutamic oxaloacetic transaminase (SGOT) and serum glutamate pyruvate transaminase (SGPT) =< 3 x ULN
* Absolute neutrophil count (ANC) >= 1,000 cell/mm^3 without growth factor support within 14 days prior to registration
* Platelets >= 50,000 cells/mm^3 for patients who have bone marrow plasmacytosis < 50% or >= 30,000 cells/mm^3 for patients who have bone marrow plasmacytosis of >= 50% within 14 days prior to registration
* Calculated or measured creatinine clearance >= 30 ml/min within 14 days prior to registration
* Patients who are known to be human immunodeficiency virus positive (HIV+) are eligible providing they meet all of the following additional criteria within 28 days prior to registration:

  * Cluster of differentiation (CD)4 cells >= 500/mm^3
  * Viral load of < 50 copies HIV messenger ribonucleic acid (mRNA)/mm^3 if on combination antiretroviral therapy (cART) or < 25,000 copies HIV mRNA if not on cART
  * No zidovudine or stavudine as part of cART
  * Patients who are HIV+ and do not meet all of these criteria are not eligible for this study
* Patients with known hepatitis B or hepatitis C infection must have viral load < 800,000 IU/L within 28 days prior to registration
* Patients must have baseline skeletal survey to document lytic lesions, osteopenia or compression fracture within 28 days prior to registration
* Patients may have received palliative external beam radiation therapy (XRT) for local disease control with no curative intent. XRT must be completed at least 7 days prior to registration
* Patients must be offered participation in specimen submission for translational medicine studies and banking; with patient consent, specimens must be submitted
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years
* Patients or their legally authorized representative must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system
* REGISTRATION STEP 2: CROSSOVER
* Patient must have been eligible for and initially randomized to Arm 1 (low dose carfilzomib), begun cycle 2 of treatment, and progressed prior to completing 12 cycles of protocol therapy
* At least 14 days and no more than 28 days must have elapsed between the last day of treatment on Arm 1 and registration to Arm 3
* Patients must have recovered from all non-hematologic toxicities to =< grade 2 and from all hematologic toxicities to =< grade 3 prior to registration
* Patients must have begun cycle 2 (carfilzomib - 27 mg/m^2) and must not have received any dose reduction for toxicity in the last cycle of treatment, immediately preceding progression
* Patients must have serum protein electrophoresis (SPEP) and kappa and lambda light chain testing performed within 14 days prior to registration in order to establish baseline measurements
* Patients must not have ejection fraction decrease > 10% from baseline (as determined by ECHO) or other ejection fraction decrease accompanied by other clinical signs/symptoms of New York Heart Association (NYHA) class III or IV heart failure, measured within 28 days prior to registration; if any question exists regarding individual patient eligibility in this situation, contact the study chair for determination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2013-10; Primary Completion 2017-11-21 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sikander Ailawadhi, Principal Investigator — SWOG Cancer Research Network
Locations (485):
- United States (485):
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - The University of Arizona Medical Center-University Campus, Tucson, Arizona
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - John Muir Medical Center-Concord Campus, Concord, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente Hospital, Fontana, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Kaiser Permanente, Fresno, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Los Angeles County-USC Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Memorial Medical Center, Modesto, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Sutter Cancer Research Consortium, Novato, California
  - Kaiser Permanente-Oakland, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter General Hospital, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - Kaiser Permanente, Woodland Hills, California
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Medical Oncology and Hematology Group PC-Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Charlotte Hungerford Hospital Center for Cancer Care, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Gynecologic Oncology LLC, Newark, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Castle Medical Center, Kailua, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Center of Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Hematology Oncology Associates-Quad Cities, Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita NCI Community Oncology Research Program, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Hematology/Oncology Clinic LLP, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Medical Oncology LLC, Baton Rouge, Louisiana
  - Mary Bird Cancer Center/Saint Tammany Parish, Covington, Louisiana
  - Mary Bird Perkins Cancer Center/Terrebonne General Medical Center, Houma, Louisiana
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Beverly Hospital, Beverly, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Providence Hospital-Southfield Cancer Center, Southfield, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro Minnesota Community Oncology Research Consortium, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Central Care Cancer Center-Carrie J Babb Cancer Center, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - CoxHealth Cancer Center, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Saint John's Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Cancer Research for the Ozarks NCORP, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Montana Cancer Consortium NCORP, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology - Fort Apache, Las Vegas, Nevada
  - Cancer and Blood Specialists-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - 21st Century Oncology - Vegas Tenaya, Las Vegas, Nevada
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - Orange Regional Medical Center, Middletown, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Cone Health Cancer Center at Alamance Regional, Burlington, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Cone Heath Cancer Center at Mebane, Mebane, North Carolina
  - Annie Penn Memorial Hospital, Reidsville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus NCI Community Oncology Research Program, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton NCI Community Oncology Research Program, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lancaster Radiation Oncology, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - OneHealth Marion General Hospital, Marion, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Wright-Patterson Medical Center, Wright-Patterson Air Force Base, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazleton, Hazleton, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Geisinger Medical Oncology-Pottsville, Pottsville, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Main Line Health NCORP, Wynnewood, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - M D Anderson Cancer Center, Houston, Texas
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Pacific Medical Center-First Hill, Seattle, Washington
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Saint Mary's Hospital, Rhinelander, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Marshfield Clinic Cancer Care at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - ProHealth Waukesha Memorial Hospital, Waukesha, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Ailawadhi S, Sexton R, Lentzsch S, Abidi MH, Voorhees PM, Cohen AD, Rohren EM, Heitner S, Kelly K, Mackler NJ, Baer DM, Hoering A, Durie B, Orlowski RZ. Low-dose versus High-dose Carfilzomib with Dexamethasone (S1304) in Patients with Relapsed-Refractory Multiple Myeloma. Clin Cancer Res. 2020 Aug 1;26(15):3969-3978. doi: 10.1158/1078-0432.CCR-19-1997. Epub 2020 Apr 16. PMID 32299820

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Dexamethasone, Low-dose Carfilzomib) | Arm II (Dexamethasone, High-dose Carfilzomib)
Started | 72 | 71
Crossover to Arm II | 16 (Following disease progression on Arm I. Note: these patients are also counted in 'Completed'.) | 0
Completed (Completed implies patients were eligible for study treatment and analyzable for study endpoints.) | 64 | 57
Not Completed | 8 | 14
Not completed — No measurable disease | 1 | 1
Not completed — Incomplete/discontinued prior therapy | 1 | 1
Not completed — Baseline lab missing/incomplete/untimely | 6 | 11
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Includes patients who were eligible and analyzable for study endpoints (indicated as "Completed" in participant flow).
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Dexamethasone, Low-dose Carfilzomib) | Arm II (Dexamethasone, High-dose Carfilzomib) | Total
Number analyzed (Participants) | 64 | 57 | 121
Age, Customized [Count of Participants; unit: Participants]
  Age >= 65 | 31 | 32 | 63
  Age < 65 | 33 | 25 | 58
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 24 | 55
  Male | 33 | 33 | 66
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 51 | 41 | 92
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 3 | 3
Zubrod performance status > 1 [Count of Participants; unit: Participants] — POINT DESCRIPTION 0: Fully active, able to carry on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of limited self-care, confined to bed or chair more than 50% of waking hours.
  4. Completely disabled; cannot carry on any self-care; totally confined to bed or chair.
  Participants | 2 | 3 | 5
Beta-2-microglobulin >=3.5 mg/L [Count of Participants; unit: Participants] | 36 | 31 | 67
CRP >= 8 mg/L [Count of Participants; unit: Participants] — Population: Due to missing/not done labs, number analyzed in row differs from overall.
  Participants
    number analyzed (Participants) | 33 | 23 | 56
    (all) | 6 | 6 | 12
Creatinine >= 2 mg/dl [Count of Participants; unit: Participants] | 1 | 0 | 1
Creatinine clearance < 60 ml/min [Count of Participants; unit: Participants] | 23 | 18 | 41
LDH >= 190 U/L [Count of Participants; unit: Participants] — Population: Due to missing/not done labs, number analyzed in row differs from overall.
  Participants
    number analyzed (Participants) | 63 | 56 | 119
    (all) | 31 | 26 | 57
Albumin < 3.5 g/dl [Count of Participants; unit: Participants] | 16 | 14 | 30
ISS disease stage: Stage 1 [Count of Participants; unit: Participants] — Stage Criteria:
  I: Serum β2-microglobulin < 3.5 mg/L Serum albumin ≥ 3.5 g/dL II: Not Stage I or III III: Serum β2-microglobulin > 5.5 mg/L
  Note: Expected survival outcomes worsen with increasing stage.
  Participants | 20 | 22 | 42
ISS disease stage: Stage 2 [Count of Participants; unit: Participants] — Stage Criteria:
  I: Serum β2-microglobulin < 3.5 mg/L Serum albumin ≥ 3.5 g/dL II: Not Stage I or III III: Serum β2-microglobulin > 5.5 mg/L
  Note: Expected survival outcomes worsen with increasing stage.
  Participants | 30 | 19 | 49
ISS disease stage: Stage 3 [Count of Participants; unit: Participants] — Stage Criteria:
  I: Serum β2-microglobulin < 3.5 mg/L Serum albumin ≥ 3.5 g/dL II: Not Stage I or III III: Serum β2-microglobulin > 5.5 mg/L
  Note: Expected survival outcomes worsen with increasing stage.
  Participants | 14 | 16 | 30
Hemoglobin <10 g/dL [Count of Participants; unit: Participants] | 15 | 6 | 21
Platelet count < 150 x 10^9/L [Count of Participants; unit: Participants] | 1 | 1 | 2
4-6 Prior lines of therapy [Count of Participants; unit: Participants] | 14 | 15 | 29
Refractory to Bortezomib [Count of Participants; unit: Participants] | 32 | 28 | 60
Serum M spike >3 g/dL [Count of Participants; unit: Participants] — Population: Due to missing/not done labs, number analyzed in row differs from overall.
  Participants
    number analyzed (Participants) | 64 | 56 | 120
    (all) | 13 | 6 | 19
Bone marrow plasma cells > 60% [Count of Participants; unit: Participants] — Population: Due to missing/not done labs, number analyzed in row differs from overall.
  Participants
    number analyzed (Participants) | 63 | 56 | 119
    (all) | 14 | 11 | 25
sLFC Ratio >=100 [Count of Participants; unit: Participants] — Population: Due to missing/not done labs, number analyzed in row differs from overall.
  Participants
    number analyzed (Participants) | 60 | 51 | 111
    (all) | 24 | 19 | 43
Myeloma isotype: IgG [Count of Participants; unit: Participants] — Population: Due to missing/not done labs, number analyzed in row differs from overall.
  Participants
    number analyzed (Participants) | 61 | 54 | 115
    (all) | 36 | 24 | 60
Myeloma isotype: IgA [Count of Participants; unit: Participants] — Population: Due to missing/not done labs, number analyzed in row differs from overall.
  Participants
    number analyzed (Participants) | 61 | 54 | 115
    (all) | 5 | 12 | 17
Myeloma isotype: light chain only [Count of Participants; unit: Participants] — Population: Due to missing/not done labs, number analyzed in row differs from overall.
  Participants
    number analyzed (Participants) | 61 | 54 | 115
    (all) | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Assessed in each arm using the method of Kaplan Meier and compared between arms using the stratified long-rank test. Progression is defined using the International Uniform Response Criteria for Multiple Myeloma as new or increase in size of existing bone lesions or soft tissue plasmacytomas; or development of hypercalcemia attributable solely to MM; or ≥ 25% increase from baseline or lowest response level of either serum M protein, urine M protein, difference in involved & uninvolved serum free light chain level or bone marrow plasma cell percentage.
Time Frame: From date of registration to date of first documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 2 years
Population: Group of participants that were eligible and analyzable per protocol.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm I (Dexamethasone, Low-dose Carfilzomib): Patients receive 20 mg dexamethasone IV and low-dose (27 mg/m^2) carfilzomib IV over 2-10 minutes on days 1, 2, 8, 9, 15, and 16. (Note that course 1 is given at a reduced dose of 20 mg/m^2.) Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity. Patients with progression cross-over to Arm II.
  Carfilzomib: Given IV
  Dexamethasone: Given IV
  Laboratory Biomarker Analysis: Correlative studies
- Arm II (Dexamethasone, High-dose Carfilzomib): Patients receive 20 mg dexamethasone IV and high-dose (56 mg/m^2) carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16. (Note that course 1 is given at a reduced dose of 20 mg/m^2 over 2-10 minutes.) Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Carfilzomib: Given IV
  Dexamethasone: Given IV
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Arm I (Dexamethasone, Low-dose Carfilzomib) | Arm II (Dexamethasone, High-dose Carfilzomib)
Number analyzed (Participants) | 64 | 57
months | 5 [4 to 11] | 8 [6 to 12]
Statistical Analysis 1: Comparison: Arm I (Dexamethasone, Low-dose Carfilzomib) vs Arm II (Dexamethasone, High-dose Carfilzomib); Test type: Superiority; p = 0.384, Log Rank — Stratified by pre-specified randomization stratification factors: 1 - 3 prior therapies vs. 4-6 prior therapies and refractory to bortezomib vs. not refractory to bortezomib; One-sided stratified log rank test; Hazard Ratio (HR) = 1.061, 80% CI 2-sided [0.821 to 1.370]

2. Secondary Outcome: Overall Survival
Description: Assessed in each arm using the method of Kaplan Meier and compared between arms using the stratified log-rank test.
Time Frame: From date of registration to date of death due to any cause, assessed up to 3 years
Population: Participants that were eligible and analyzable per protocol.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Dexamethasone, Low-dose Carfilzomib) | Arm II (Dexamethasone, High-dose Carfilzomib)
Number analyzed (Participants) | 64 | 57
months | 26 [16 to NA] — The upper limit for this 95% confidence interval for the median is not calculable. | 22 [18 to 29]
Statistical Analysis 1: Comparison: Arm I (Dexamethasone, Low-dose Carfilzomib) vs Arm II (Dexamethasone, High-dose Carfilzomib); Test type: Superiority; p = 0.284, Log Rank — [p-value comment as in outcome 1, analysis 1]; One-sided stratified log rank test; Hazard Ratio (HR) = 1.149, 80% CI 2-sided [0.841 to 1.571]

3. Secondary Outcome: Best Overall Response - Partial Response (PR), Very Good Partial Response (VGPR), Unconfirmed PR (uPR), Stable Disease (SD) Progression (PROG)
Description: Per International Uniform Response Criteria for Multiple Myeloma PR- ≥ 50% reduction in size of soft tissue plasmacytomas & plasma cells; ≥ 50% decrease in serum & reduction in urine M protein ≥ 90% or to < 200 mg/24hr or ≥ 50% decrease in difference in uninvolved & involved serum free light chain levels; VGPR- PR + Serum and urine M proteins detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M protein & urine M protein < 100 mg/24 hrs; uPR- 1 objective status of PR, but confirmation studies are not done, or do not meet the requirements necessary to confirm response; SD- does not meet criteria for sCR, CR, VGPR, PR or PROG; PROG- new or increase in size of existing bone lesions or soft tissue plasmacytomas/ development of hypercalcemia attributable solely to MM/ ≥ 25% increase from baseline/ lowest response level of either serum or Urine M protein, difference in involved & uninvolved serum free light chain level or bone marrow plasma cell percentage.
Time Frame: From date of registration to date of best response while on study treatment
Population: This population includes eligible and analyzable patients who had a follow-up response assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Dexamethasone, Low-dose Carfilzomib) | Arm II (Dexamethasone, High-dose Carfilzomib)
Number analyzed (Participants) | 59 | 53
Participants
  Very Good Partial Response (VGPR) | 5 | 14
  Partial Response (PR) | 18 | 11
  Unconfirmed Partial Response (uPR) | 0 | 2
  Stable Disease (SD) | 24 | 19
  Progressive Disease | 12 | 7
Statistical Analysis 1: Comparison: Arm I (Dexamethasone, Low-dose Carfilzomib) vs Arm II (Dexamethasone, High-dose Carfilzomib); Compare the rate of confirmed PR or better between treatment arms; Test type: Superiority; p = 0.1130, Cochran-Mantel-Haenszel

4. Secondary Outcome: Progression-free Survival of Crossover Group
Description: Assessed in the crossover arm using the method of Kaplan Meier. Progression is defined using the International Uniform Response Criteria for Multiple Myeloma as new or increase in size of existing bone lesions or soft tissue plasmacytomas; or development of hypercalcemia attributable solely to MM; or ≥ 25% increase from baseline or lowest response level of either serum M protein, urine M protein, difference in involved & uninvolved serum free light chain level or bone marrow plasma cell percentage.
Time Frame: From date of crossover to date of subsequent documentation of progression or symptomatic deterioration, or death due to any cause, assessed up to 3 years from randomization
Population: Patients on Arm 1 that progress after the start of course 2 and prior to completion of 12 courses receive high dose carfilzomib
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm III (Crossover Group): Patients on Arm 1 that progress after the start of course 2 and prior to completion of 12 courses receive 20 mg dexamethasone IV and high-dose (56 mg/m^2) carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for up to 12 additional courses in the absence of disease progression or unacceptable toxicity.
  Carfilzomib: Given IV Dexamethasone: Given IV Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Arm III (Crossover Group)
Number analyzed (Participants) | 16
months | 3 [2 to 6]

5. Secondary Outcome: Overall Survival Crossover Group
Description: Assessed in the crossover arm using the method of Kaplan Meier.
Time Frame: From date of crossover to date of death due to any cause, assessed up to 3 years from randomization
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Crossover Arm: Patients on Arm 1 that progress after the start of course 2 and prior to completion of 12 courses receive 20 mg dexamethasone IV and high-dose (56 mg/m^2) carfilzomib IV over 30 minutes on days 1, 2, 8, 9, 15, and 16. Treatment repeats every 28 days for up to 12 additional courses in the absence of disease progression or unacceptable toxicity.
  Carfilzomib: Given IV Dexamethasone: Given IV Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Crossover Arm
Number analyzed (Participants) | 16
months | 15 [5 to 27]

6. Other Pre Specified Outcome: Gene Expression Profiles
Description: Bone marrow compared to that of an aspirate taken at the site of the EMP. Data will be log-transformed before analysis. Exploratory analyses will examine underlying distributions using boxplots, density plots, scatter plots, etc. For differential expression analysis of the two sample types t-tests will be conducted on genes. False discovery rate will be used to control the average false positive proportions among selected genes. Genes will be ranked by their q-value and pathway analysis conducted upon selected genes to determine biological plausibility and relevance to molecular functionality.
Time Frame: Up to 3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Incidence of CR by PET, Defined as the Disappearance of All Focal Lesions and the Resolution of EMD
Description: Univariate and multivariate logistic regression will be used to determine the impact of biochemical CR on CR by PET. In the multivariate analysis adjustment for standard prognostic factors such as age, albumin, beta-2 microglobulin, serum creatinine, c-reactive protein and lactate dehydrogenase will be included.
Time Frame: Up to week 45
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: For the duration of treatment, up to 12 cycles and maximum follow up of 3 years post-registration.
Description: Note that denominators differ from those reported in other Results sections as the AE data tables are pulled from the live database and thus reflect more current data while other Sections are based those data reported at the time of Primary Endpoint analyses.
Groups:
- Arm I (Dexamethasone, Low-dose Carfilzomib): Patients receive dexamethasone and low dose carfilzomib. Includes all eligible and analyzable patients. Deaths for patients that registered Crossover arm are also counted in this arm.
- Arm II (Dexamethasone, High-dose Carfilzomib): Patients receive dexamethasone and high dose carfilzomib. Includes all eligible and analyzable patients.
- Crossover Arm: Patients on Arm 1 that progress after the start of cycle 2 and prior to completion of 12 cycles receive high dose carfilzomib. Includes all eligible and analyzable patients. These patients are also included under "Arm I".
Arm/Group | Arm I (Dexamethasone, Low-dose Carfilzomib) | Arm II (Dexamethasone, High-dose Carfilzomib) | Crossover Arm
All-Cause Mortality (participants affected / at risk) | 38/66 | 40/57 | 12/16
Serious Adverse Events (participants affected / at risk) | 26/66 | 27/57 | 5/16
Other Adverse Events (participants affected / at risk) | 66/66 | 55/57 | 14/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Dexamethasone, Low-dose Carfilzomib) (N=66) | Arm II (Dexamethasone, High-dose Carfilzomib) (N=57) | Crossover Arm (N=16)
Anemia (Blood and lymphatic system disorders) | 3 | 6 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0
Heart failure (Cardiac disorders) | 2 | 2 | 0
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 2 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Blurred vision (Eye disorders) | 2 | 0 | 0
Glaucoma (Eye disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0
Chills (General disorders) | 0 | 1 | 0
Death NOS (General disorders) | 1 | 1 | 0
Edema limbs (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 2 | 3 | 0
Fever (General disorders) | 2 | 6 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Sudden death NOS (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Endocarditis infective (Infections and infestations) | 0 | 1 | 0
Infections and infestations-Other (Infections and infestations) | 2 | 0 | 0
Lung infection (Infections and infestations) | 3 | 7 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 2 | 3 | 2
Sinusitis (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 0 | 0
Creatinine increased (Investigations) | 2 | 2 | 0
Ejection fraction decreased (Investigations) | 2 | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 3 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 4 | 7 | 1
White blood cell decreased (Investigations) | 1 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Nervous system disorders-Other (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Stroke (Nervous system disorders) | 0 | 2 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Confusion (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 0 | 2 | 0
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 | 1 | 0
Renal calculi (Renal and urinary disorders) | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Hypotension (Vascular disorders) | 2 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Dexamethasone, Low-dose Carfilzomib) (N=66) | Arm II (Dexamethasone, High-dose Carfilzomib) (N=57) | Crossover Arm (N=16)
Anemia (Blood and lymphatic system disorders) | 39 | 38 | 8
Cardiac disorders-Other (Cardiac disorders) | 5 | 2 | 0
Chest pain - cardiac (Cardiac disorders) | 1 | 3 | 1
Sinus bradycardia (Cardiac disorders) | 4 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 7 | 3 | 0
Hearing impaired (Ear and labyrinth disorders) | 1 | 3 | 0
Blurred vision (Eye disorders) | 9 | 11 | 0
Watering eyes (Eye disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 6 | 8 | 1
Bloating (Gastrointestinal disorders) | 0 | 4 | 0
Constipation (Gastrointestinal disorders) | 12 | 14 | 2
Diarrhea (Gastrointestinal disorders) | 20 | 20 | 2
Dry mouth (Gastrointestinal disorders) | 6 | 7 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 7 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 4 | 4 | 0
Nausea (Gastrointestinal disorders) | 25 | 21 | 5
Stomach pain (Gastrointestinal disorders) | 2 | 3 | 2
Vomiting (Gastrointestinal disorders) | 13 | 9 | 0
Chills (General disorders) | 5 | 5 | 2
Edema face (General disorders) | 5 | 1 | 1
Edema limbs (General disorders) | 14 | 9 | 1
Fatigue (General disorders) | 39 | 33 | 6
Fever (General disorders) | 9 | 5 | 2
Flu like symptoms (General disorders) | 5 | 2 | 1
Non-cardiac chest pain (General disorders) | 4 | 4 | 0
Pain (General disorders) | 13 | 15 | 1
Allergic reaction (Immune system disorders) | 0 | 0 | 1
Immune system disorders-Other (Immune system disorders) | 1 | 1 | 1
Infections and infestations-Other (Infections and infestations) | 5 | 6 | 0
Sinusitis (Infections and infestations) | 5 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 1
Upper respiratory infection (Infections and infestations) | 5 | 7 | 1
Bruising (Injury, poisoning and procedural complications) | 5 | 6 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 4 | 0
Alkaline phosphatase increased (Investigations) | 7 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 7 | 8 | 0
Blood bilirubin increased (Investigations) | 8 | 4 | 0
Creatinine increased (Investigations) | 15 | 14 | 2
Lymphocyte count decreased (Investigations) | 18 | 16 | 4
Neutrophil count decreased (Investigations) | 13 | 14 | 1
Platelet count decreased (Investigations) | 28 | 29 | 5
Weight gain (Investigations) | 7 | 3 | 1
Weight loss (Investigations) | 5 | 8 | 0
White blood cell decreased (Investigations) | 21 | 24 | 3
Anorexia (Metabolism and nutrition disorders) | 12 | 13 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 6 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 4 | 2 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 15 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 5 | 2 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 5 | 4 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 | 15 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 11 | 0
Hypokalemia (Metabolism and nutrition disorders) | 13 | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 9 | 8 | 0
Hyponatremia (Metabolism and nutrition disorders) | 9 | 11 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 5 | 7 | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 11 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 21 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 6 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 | 8 | 1
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 5 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 15 | 3
Dizziness (Nervous system disorders) | 13 | 12 | 1
Dysgeusia (Nervous system disorders) | 3 | 4 | 1
Headache (Nervous system disorders) | 20 | 18 | 2
Nervous system disorders-Other (Nervous system disorders) | 1 | 3 | 0
Paresthesia (Nervous system disorders) | 5 | 4 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 5 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 20 | 18 | 4
Anxiety (Psychiatric disorders) | 10 | 9 | 2
Confusion (Psychiatric disorders) | 4 | 3 | 2
Depression (Psychiatric disorders) | 8 | 3 | 2
Insomnia (Psychiatric disorders) | 19 | 20 | 3
Acute kidney injury (Renal and urinary disorders) | 3 | 2 | 1
Chronic kidney disease (Renal and urinary disorders) | 2 | 3 | 1
Proteinuria (Renal and urinary disorders) | 6 | 2 | 0
Renal and urinary disorders-Other (Renal and urinary disorders) | 3 | 1 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 17 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 22 | 27 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8 | 7 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Flushing (Vascular disorders) | 8 | 4 | 0
Hot flashes (Vascular disorders) | 1 | 3 | 0
Hypertension (Vascular disorders) | 16 | 20 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-12-10): https://cdn.clinicaltrials.gov/large-docs/11/NCT01903811/Prot_SAP_ICF_000.pdf